CLINICAL TRIAL: NCT06930313
Title: Development and Evaluation of a Brief Compassion-Based Intervention for Managing Depression and Anxiety in Family Caregivers of Lung Cancer Patients: A Mixed Methods Randomized Controlled Trial
Brief Title: Compassion-Based Intervention for Lung Cancer Caregivers (CBI-LCC)
Acronym: CBI-LCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N202411055; IRB Approval Number (Other: TMU-Joint Institutional Review Board)
Record Dates: First submitted 2025-01-14; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-01

CONDITIONS: Compassion
Keywords: compassion-based intervention; lung cancer; family caregivers; caregiver stress; depression; anxiety; mindfulness; self-compassion
MeSH Terms: conditions — Lung Neoplasms; Caregiver Burden; Depression; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Arm 1: Experimental Arm Name: Brief Compassion-Based Intervention (BCI) Description: Participants in this arm will receive a 4-session Brief Compassion-Based Intervention (BCI) focused on managing depression and anxiety in family caregivers of lung cancer patients.
  Arm 2: Control Arm Name: Telephone-Based Support and Education (TSE) Description: Participants in this arm will receive a single-session Telephone-Based Support and Education (TSE), providing general caregiving advice and emotional support.
Who Masked: Participant, Investigator
Masking Description: Participant Masking Description: Participants will not be informed of their group allocation (Intervention or Control group). While participants will know the specific type of support they are receiving (e.g., Compassion-Based Intervention or Telephone-Based Support), they will not be aware of which group is considered the experimental intervention.
  Investigator Masking: Investigators responsible for data collection and analysis will be blinded to group allocation to maintain objectivity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Compassion-Based Intervention (BCI) (Experimental): Participants in this arm will receive a 4-session Brief Compassion-Based Intervention (BCI) focused on managing depression and anxiety in family caregivers of lung cancer patients.
  Interventions: Behavioral: Brief Compassion-Based Intervention (BCI)
- Telephone-Based Support and Education (TSE) (Active Comparator): Participants in this arm will receive a single-session Telephone-Based Support and Education (TSE), providing general caregiving advice and emotional support.
  Interventions: Behavioral: Telephone-Based Support and Education (TSE)

INTERVENTIONS:
Behavioral: Brief Compassion-Based Intervention (BCI) — The intervention program is based on Compassion-Focused Therapy (CFT) and incorporates evidence-based compassion exercises.Drawing on insights from the literature, the program includes:Session 1: Introduction to caregiving challenges and emotional systems. Includes a soothing breathing exercise and group discussion on caregiving stress.
  Session 2: Cultivating self-compassion. Includes reflecting on emotions, guided meditation, and a compassionate body scan practice.
  Session 3: Transforming self-criticism into self-compassion. Caregivers explore self-critical thoughts, practice reframing, and engage in compassionate dialogue.
  Session 4: Building resilience and connections. Focuses on gratitude, setting boundaries, and loving-kindness meditation, ending with daily intention setting.
  Arms: Brief Compassion-Based Intervention (BCI)
Behavioral: Telephone-Based Support and Education (TSE) — The session will address their questions and concerns, provide psychological support for managing difficult emotions (e.g., anxiety, fear, sadness, and guilt), and emphasize the importance of self-care, encouraging them to take time for themselves and seek support when needed.
  Arms: Telephone-Based Support and Education (TSE)

SUMMARY:
Objectives: This 3-year study aims to develop, refine, and evaluate a brief compassion-based intervention specifically designed for family caregivers of lung cancer patients. In the first year, the primary focus will be on developing the intervention content and assessing its feasibility and acceptability. In the second and third years, the goal will be to assess the intervention's effects on depression and anxiety.

Method: In the first year, the intervention will be developed in three stages. Initially, the intervention will be created based on compassion-focused theory and evidence-based exercises, incorporating feedback from family caregivers in previous studies and insights from professionals to ensure its relevance to lung cancer caregivers. Next, a pilot study will test the intervention's feasibility and acceptability with 30 family caregivers, using mixed methods to gather session-by-session feedback and assess recruitment, retention, and adherence. Following the pilot, the intervention will be revised based on participant and researcher feedback, preparing it for further study. In the second and third years, a randomized controlled trial (RCT) will be conducted with 84 participants randomly assigned to either the 4-session Brief Compassion-Based Intervention (BCI) or a single-session Telephone-Based Support and Education (TSE) control group. Outcomes, including depression, anxiety, caregiver stress, mindfulness, self-compassion, and self-efficacy, will be measured at baseline, immediately post-intervention, and at 3- and 6-month follow-ups. For data analysis, long-term follow-up quantitative data will be analyzed using the Generalized Estimating Equation (GEE) to examine group differences. Moderation and mediation analyses will be conducted to explore potential moderators and mechanisms of the intervention. Qualitative data from interviews will be analyzed using content analysis.

Expected Results: This study is expected to provide a comprehensive understanding of the feasibility, acceptability, and effectiveness of compassion-based interventions for lung cancer caregivers, contributing to their application in clinical care practice.

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregiver of a person with newly diagnosed lung cancer (within one year of diagnosis)
* Aged 20 years or older
* Access to a computer or smartphone with internet connection at home

Exclusion Criteria:

* Currently receiving psychological therapy
* Diagnosed with a severe mental illness and taking medication for it (e.g.,psychosis, bipolar disorder)
* Previous experience with mindfulness or self-compassion training

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) Questionnaire | From baseline through study completion, up to 6 months.
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS), a validated self-report questionnaire developed by Zigmond and Snaith in 1983. The HADS comprises 14 items divided into two subscales: anxiety (7 items) and depression (7 items). Participants will rate the frequency of symptoms experienced during the past week on a 4-point Likert scale ranging from 0 ("not at all") to 3 ("most of the time"). Scores on each subscale range from 0 to 21, with higher scores indicating greater levels of anxiety or depression.

SECONDARY OUTCOMES:
Kingston Caregiver Stress Scale (KCSS) Questionnaire | From baseline through study completion, up to 6 months.
  Caregiving-related stress will be assessed using the Kingston Caregiver Stress Scale (KCSS), a validated self-report questionnaire developed by Sadak et al. (2017). The KCSS includes 10 items measuring caregivers' perceived stress across three domains: caregiving duties (7 items), family-related pressures (2 items), and financial challenges (1 item). Items are rated on a 5-point Likert scale ranging from 1 ("feeling fine/no stress") to 5 ("extreme stress"). Total scores range from 10 to 50, with higher scores indicating greater levels of caregiving stress.
Five Facet Mindfulness Questionnaire (FFMQ-15) | From baseline through study completion, up to 6 months.
  Mindfulness will be assessed using the 15-item Five Facet Mindfulness Questionnaire (FFMQ-15), a validated self-report questionnaire that evaluates five facets of mindfulness: observing, describing, acting with awareness, non-judgment, and non-reactivity. Participants rate their agreement with each item on a 5-point Likert scale ranging from 1 ("rarely true") to 5 ("always true"). Scores from each item are summed to produce a total mindfulness score ranging from 15 to 75, with higher scores indicating greater mindfulness.
Self-Compassion Scale (SCS) Questionnaire | From baseline through study completion, up to 6 months.
  Self-compassion will be assessed using the Self-Compassion Scale, a validated 13-item self-report questionnaire developed by Gilbert et al. (2017). This measure evaluates an individual's capacity for self-compassion across two subscales. Participants rate each item on a 10-point Likert scale ranging from 1 ("Never") to 10 ("Always"). The two subscale scores are summed to produce a total score, with higher scores indicating greater self-compassion.
General Self-Efficacy Scale (GSES) Questionnaire | From baseline through study completion, up to 6 months.
  Self-efficacy will be assessed using the General Self-Efficacy Scale (GSES), a validated 10-item self-report questionnaire developed by Schwarzer and Jerusalem (1995). The GSES evaluates an individual's perception of their capability to manage daily challenges and cope effectively with stressful life events. Participants rate each item on a 4-point Likert scale ranging from 1 ("not at all") to 4 ("exactly true"). Total scores range from 10 to 40, with higher scores indicating greater self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan, Taiwan